CLINICAL TRIAL: NCT04086030
Title: Postoperative Blood Flow Restriction Training Following Anterior Cruciate Ligament Reconstruction: A Randomized Clinical Trial.
Brief Title: Blood Flow Restriction Following ACLR
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Could not recruit participants for study
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19050802
Record Dates: First submitted 2019-09-04; First posted 2019-09-11 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Anterior Cruciate Ligament Injuries; ACL; Physical Therapy
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham Postoperative Rehabilitation (Sham Comparator): Patients in this group will complete the standardized postoperative rehabilitation program with sham BFR, which is pressure of 20 mmHG. Exercises will be performed for 4 sets of 30/15/15/15 repetitions with a 30 second rest period between each set. The tourniquet cuff will remain inflated for all sets and rest periods for the selected exercise. A cadence of 2-second concentric and 2- second eccentric contractions (4 second time under tension) will be maintained for each BFR repetition. Upon completion of the exercise, the tourniquet cuff will be deflated, and a 1 minute minimum rest period will occur before moving on to another BFR exercise.
  Interventions: Other: Sham Blood Flow Restriction Training
- BFR Postoperative Rehabilitation (Experimental): Assigned intervention of BFR where exercises are performed with BFR at 80% limb occlusion pressure (LOP). Patients in this group will undergo blood flow restriction (BFR) training during their postoperative rehabilitation program (use an inflatable cuff that prevents blood flow from flowing out of the leg while patients perform physical therapy exercises). Exercises will be performed for 4 sets of 30/15/15/15 repetitions with a 30 second rest period between each set.16 The tourniquet cuff will remain inflated for all sets and rest periods for the selected exercise. A cadence of 2-second concentric and 2- second eccentric contractions (4 second time under tension) will be maintained for each BFR repetition. Upon completion of the exercise, the tourniquet cuff will be deflated, and a 1 minute minimum rest period will occur before moving on to another BFR exercise.
  Interventions: Other: Blood Flow Restriction Training

INTERVENTIONS:
Other: Blood Flow Restriction Training — Patients will undergo standardized postoperative rehabilitation program including blood flow restriction training. Exercises will be performed with BFR at 80% LOP.
  Arms: BFR Postoperative Rehabilitation
Other: Sham Blood Flow Restriction Training — Patients will undergo standardized postoperative rehabilitation program where exercises will be performed with sham BFR pressure of 20 mmHG.
  Arms: Sham Postoperative Rehabilitation

SUMMARY:
The purpose of this study is to evaluate the the ability of BFR to reduce muscle loss and improve strength after ACL reconstruction. It is hypothesized that BFR training will significantly reduce muscle loss and improve strength after ACL reconstruction. It is also hypothesized that BFR will result in improved patient reported outcomes and rates of return to sport.

DETAILED DESCRIPTION:
Following anterior cruciate ligament (ACL) reconstruction, many patients experience weakness of the quadriceps (thigh muscles) and loss of muscle mass due to inactivity following surgery. Recent research has demonstrated that blood flow restriction (BFR) training can help reduce the loss of muscle mass and strength after surgery. Blood flow restriction training uses an inflatable cuff that prevents blood from flowing out of the leg while patients perform physical therapy exercises. This allows patients to use lighter weights while reducing muscle loss and building strength.

This will be a prospective, randomized controlled trial of patients undergoing ACL reconstruction with bone-patellar tendon-bone (BTB) autograft. Half the subjects will be randomly assigned to the BFR group and half will undergo sham BFR therapy after surgery.

Statistical Assumptions: To sufficiently power (80%) the investigation to detect a difference (alpha = 0.05) in quadriceps muscle strength (isokinetic contraction) following the completion of the BFR rehabilitation program, 19 subjects per group (38 total) would be required. However, accounting for a 20% attrition rate and an additional 20% potentially screened out at the time of surgery due to other pathology (i.e. repairable meniscus tears, cartilage defects, etc.) that alters the prescribed physical therapy protocol, this study will aim to recruit and enroll 54 subjects (27 per group).

Following ACL reconstruction surgery, subjects will complete a standardized postoperative rehabilitation program with or without BFR. The rehabilitation program will be broken into 4 phases including (1) protection, range of motion, and proprioception; (2) strength and endurance; (3) power and agility; and (4) return to sport training. Physical therapy will occur 2 times per week for 20 weeks. Subjects will attend follow-up visits at 1, 3, 6, and 12 months. Physical exam and muscle mass measurements will be performed at all visits, while strength testing will be performed at 3, 6, and 12 months.

The goal of this study is to determine the efficacy of BFR therapy in improving muscle strength and reducing loss of muscle mass following ACL reconstruction, in addition to determining the effect of BFR on patient reported outcomes and return to sport. It is anticipated that BFR will significantly reduce the loss of muscle mass and improve muscular strength compared to standard therapy. It is also expected that these subjects will have improved patient reported outcomes and greater rates of return to sport.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18-40
* English-speaking
* Primary ACL Reconstruction
* No associated procedures (meniscal repair, other ligamentous pathology), or history of deep vein thrombosis.
* Clinical and radiographic examination (MRI) consistent with an acute full thickness ACL tear and surgical consent for ACL reconstruction with a patellar tendon autograft
* Written and informed consent for study participation

Exclusion Criteria:

* Patients younger than 18 or older than 40 years of age
* Non-native English speaker
* Revision surgery or prior history of knee surgery
* Concomitant ligamentous, meniscal, or cartilage injury that would alter postoperative weight bearing status or rehabilitation protocol
* Inability to comply with the proposed follow-up clinic visits
* Patients lacking decisional capacity
* Patients with a history of deep vein thrombosis, pulmonary embolism, or known clotting disorder or hypercoagulable state
* Pregnant or breast-feeding women. Pregnancy as determined by a positive pregnancy test prior to procedure. Females of childbearing potential must agree to use an acceptable birth control method during study participation.
* Worker's compensation patients
* Any clinically significant finding that would place the patient at health risk, impact the study, or affect the completion of the study
* Any psychiatric illness that would prevent comprehension of the details and nature of the study and interfere with follow-up clinic visits

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Muscle strength | 3 month follow-up
  Quadriceps strength measured with dynamometer
Muscle strength | 6 month follow-up
  Quadriceps strength measured with dynamometer
Muscle strength | 12 month follow-up
  Quadriceps strength measured with dynamometer
Quadriceps hypertrophy | 3 month follow-up
  Standardized circumferential leg measurements to assess quadriceps hypertrophy
Quadriceps hypertrophy | 6 month follow-up
  Standardized circumferential leg measurements to assess quadriceps hypertrophy
Quadriceps hypertrophy | 12 month follow-up
  Standardized circumferential leg measurements to assess quadriceps hypertrophy